CLINICAL TRIAL: NCT06553703
Title: Effect of Acceptance and Commitment Therapy Based Group Psychoeducatıon Applied to Nursing Students on Psychological Flexibility and Somatic Symptoms
Brief Title: Acceptance and Commitment Therapy Based Group Psychoeducation for Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tugba Yildirim (Other)
Responsible Party: Sponsor-Investigator, Tugba Yildirim, Research Assistant, Çankırı Karatekin University
Organization: Çankırı Karatekin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Tuğba YILDIRIM
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-08

CONDITIONS: Psychological Flexibility; Somatic Symptom
Keywords: acceptance and commitment therapy; psychoeducation; nursing students; psychological flexibility; somatic symptom
MeSH Terms: conditions — Medically Unexplained Symptoms

STUDY DESIGN:
Intervention Model Description: In the study, 54 students were taken as sampling, 27 of which were experimental and 27 were control.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, it is not possible to blind the researcher implementing the intervention and the participants. To prevent bias in the study, the pretest will be applied before randomization. It is planned to blind the statistical and report writing process in the study. The assignment of students to the intervention and control groups will be made by a statistician independent of the study. The researcher and students will not know which group they are in until the application begins. After applying the follow-up tests, the researcher will code the data as A and B groups and transfer it to SPSS. With this method, it is planned that the statistician will do the analysis and reporting without knowing which group is the intervention and which group is the control group. It is planned to explain the codes of the groups after the analysis and reporting of the data. In this way, detection bias, statistical bias, and reporting bias will be prevented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acceptance and commitment therapy based group psychoeducation (Experimental): Acceptance and commitment therapybased group psychoeducation to be carried out with the experimental group is planned as 8 sessions. The sessions are planned to be held in 3 groups of 9 people each. The duration of a session is planned to be approximately 90 minutes. Group psychoeducation with the experimental group will be carried out face-to-face every week. The appropriate day for the sessions will be decided together with themembers of each group. The same group session will be held on the same day and time every week.
  Interventions: Other: Acceptance and commitment therapy based group psychoeducation
- No Intervention: Waiting list group (No Intervention): After the follow-up tests were completed, it was planned to apply the 8-session group psychoeducation applied to the intervention group in the same way to the control group, upon their request.
  Intervention: Acceptance and commitment therapy-based group psychoeducation aimed at increasing students' psychological flexibility and reducing their somatic symptoms.

INTERVENTIONS:
Other: Acceptance and commitment therapy based group psychoeducation — Acceptance and commitment therapy-based group psychoeducation aimed at increasing nursing students' psychological flexibility and reducing their somatic symptoms.
  Arms: Acceptance and commitment therapy based group psychoeducation

SUMMARY:
In this study, the effects of acceptance and commitment therapy-based group psychoeducation applied to nursing students on psychological flexibility and somatic symptoms will be examined. The research will be carried out as a randomized controlled experimental study with a pre-test-post-test and follow-up design.

DETAILED DESCRIPTION:
The stress factors that nursing students encounter differ from other students. One of the reasons for this is that the nursing curriculum includes working simultaneously in both theoretical and clinical environments. In a study, it was determined that nursing students' lack of stress coping skills caused internal stressors to turn into external stressors. When these individuals cannot cope with situations that cause stress, they can express the stress they experience with somatic symptoms. Somatic symptom disorder is defined as the state of seeking help for mental problems with somatic symptoms. The inability to treat these somatic symptoms of individuals forces them to live with these symptoms for years and sometimes for a lifetime and continue to seek treatment. Acceptance and Commitment Therapy, which provides a new perspective for individuals to cope with stressful life events, aims to gain psychological flexibility, which is the capacity for individuals to experience challenging conditions at the moment they are in and to behave in a way that is compatible with their value areas under these conditions. The opposite of psychological flexibility is psychological inflexibility. Experiential avoidance is one of the basic components of the concept of psychological inflexibility. The state of escape and avoidance and actions that occur when an individual does not want to be in contact with situations that stress them are defined as experiential avoidance. When the relevant literature is examined, it has been reported that somatic symptoms are seen as experiential avoidance behaviors in individuals. The continuity of somatic symptoms as a reaction to stress, their inability to intervene, and their chronicity cause them to turn into a somatic somatic symptom disorder. Since nursing students are a highly stressed group, their reactions to stress should be observed, somatic symptoms in these students should be evaluated, and psychological flexibility should be increased before somatic symptoms turn into disorders and students start their professions, and healthier members of the profession should be trained in terms of mental and physical health. However, psychosocial intervention studies that will help with somatic symptoms continue to be the subject of very little research.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* No problems understanding and speaking Turkish
* Having moderate and high-level somatic symptoms (Scoring 26 or higher on the Bradford Somatic Inventory)

Exclusion Criteria:

* Scoring 25 or less on the Bradford Somatic Inventory
* Having been diagnosed with a chronic/systemic physical illness
* Having been diagnosed with a psychiatric illness
* Being on medication for a current physical or psychiatric illness
* Have received or are receiving individual or group psychotherapy/counseling programs within the last two years
* Being a foreign national
* Being pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Change in the Psychological Flexibility Scale | Baseline, 8th week, 1st month follow-up, 3rd month follow-up) (Pretest-posttest follow-up experimental design
  The Psychological Flexibility Scale consists of 28 items and five sub-dimensions. The sub-dimensions of the scale are: "Values and committed action", "Contact with the present moment", "Acceptance", "Self as Context" and "Defusion." The increase in the scores obtained from the sub-dimensions and total scores of the scale means that individuals are psychologically flexible. The lowest score that can be obtained from the scale is 28, and the highest is 196.

SECONDARY OUTCOMES:
Bradford Somatic Symptom Inventory Change | screening, baseline, 8th week, 1st month follow-up, 3rd month follow-up) (Pretest-posttest follow-up experimental design)
  Bradford Somatic Inventory consists of 44 items. It questions the individual's experience of a wide variety of somatic symptoms on less than 15 days or more than 15 days during the previous month. In the total score of the scale, 0-25 is the low range, 26-40 is the medium range, and>40 is the high range.

OTHER OUTCOMES:
Inclusion Form | screening
  The inclusion form is a seven-question form prepared by the researcher to determine the disease status of nursing students (physical and psychiatric disease diagnosis, treatment, psychotherapy, or psychological counseling status) and sociodemographic characteristics (nationality and pregnancy status).
Participant Information Form | baseline, 8th week, 1st month follow-up, 3rd month follow-up) (Pretest-posttest follow-up experimental design)
  The participant information form is a ten-question form prepared by the researcher to determine the sociodemographic characteristics of nursing students (age, gender, class information, marital status, mother's education status, father's education status, family income status, family type, where they lived before starting university and who they currently live with).

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba YILDIRIM, Principal Investigator — Cankiri Karatekin University, Cankiri, Turkey, 18200
Locations (1):
- Tuğba Yildirim, Merkez, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Üzar Özçetin, Y.S. (2020).Somatik belirti bozukluğu ve ilişkili bozukluklar ve hemşirelik bakımı. (Ed: Akgün Çıtak E, Hiçdurmaz, D). Psikiyatri Hemşireliği Akıl Notları. 1. Baskı. Ankara: Güneş Tıp Kitabevleri. s:229-245.
- [Background] Towsend, M. (2016). Ruh Sağlığı ve Psikiyatri Hemşireliğinin Temelleri Kanıta Dayalı Uygulama Bakım Kavramları. (Çev.Ed: Tangül Özcan, C., Gürhan, N.) Ankara: Akademisyen Kitabevi. 6. Baskı. s: 516-544.
- [Background] Köse,S.,Tekintas, N.S., Durmus,F. B., Akın,E., & Sayar, K. (2017). Reliability, validity,and factorial structure of the Turkish version of the Bradford Somatic Inventory (Turkish BSI-44) in a university student sample. Psychiatry and Clinical Psychopharmacology, 27(1), 62-69.
- [Background] Kotan, Z. (2021).Somatik belirti bozukluğu ve ilişkili bozukluklarda grup terapileri. Coşar B, editör. (Ed: Coşar, B.) Somatik Belirti ve İlişkili Bozukluklar. 1. Baskı. Ankara: Türkiye Klinikleri. s: 68-73.
- [Background] Kabadayı Şahin, E. (2017). Bedensel belirti bozukluğu ve oksidatif stres. Yıldırım Beyazıt Üniversitesi Tıp Fakültesi Ruh Sağlığı ve Hastalıkları Ana Bilim Dalı Tıpta Uzmanlık tezi, Ankara.
- [Background] Ishizu K, Shimoda Y, Ohtsuki T. The reciprocal relations between experiential avoidance, school stressor, and psychological stress response among Japanese adolescents. PLoS One. 2017 Nov 22;12(11):e0188368. doi: 10.1371/journal.pone.0188368. eCollection 2017. PMID 29166647
- [Background] Hayes,S.C. (2004). Acceptanceand commitment therapy, relational frametheory and thethird wave of bahavioral and cognitivetherapies. Behavior Therapy, 35, 639-665
- [Background] Hartman,T., Blankenstein. N., Molenaar. B., & Al.E. N.H.G.(2013). Guideline on medically unexplained symptoms (MUS). Huisarts Wet, 56(5):2-18.
- [Background] Crary P. Beliefs, behaviors, and health of undergraduate nursing students. Holist Nurs Pract. 2013 Mar-Apr;27(2):74-88. doi: 10.1097/HNP.0b013e318280f75e. PMID 23399707
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Arch, J. J., & Craske, M. G. (2008). Acceptance and commitment therapy and cognitive behavioral therapy for anxiety disorders: Different treatments, similar mechanisms? Clinical Psychology: Science and Practice, 15(4), 263-279.